CLINICAL TRIAL: NCT04258605
Title: ASHCOM Shoulder System and Its Related Instruments - A Multicenter, Prospective, Non-Controlled Post Market Clinical Follow-up Study
Brief Title: ASHCOM Shoulder System and Its Related Instruments
Status: Terminated | Type: Observational
Why Stopped: Termination of PMCF study due to product discontinuation.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2017-67E
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Injuries; Shoulder Pain; Arthropathy; Traumatic; Arthroplasty Complications
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ASHCOM Shoulder System subjects: Subjects implanted with the ASHCOM Shoulder System
  Interventions: Device: ASHCOM Shoulder System

INTERVENTIONS:
Device: ASHCOM Shoulder System — Reverse Shoulder Arthroplasty

SUMMARY:
The objectives of this study are to confirm safety, performance and clinical benefits of the ASHCOM Shoulder System and its related instruments by analysis of standard scoring systems, radiographs and adverse event records.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-controlled Post-Market Clinical Follow-up study involving orthopaedic surgeons skilled in reverse shoulder arthroplasty procedures. A minimum of three study centers will be involved. A total number of 97 implants will be included into the study.

The primary endpoint is defined by the survival of the implant at 10 years which is based on removal or intended removal of the prosthesis and will be determined using Kaplan Meier method. The safety of the system will be assessed by monitoring the frequency and incidence of adverse events.

The secondary endpoint is defined by the performance and clinical benefits of the ASHCOM Shoulder System at 5 years, which is assessed by the Constant and Murley score. Assessments of the overall pain, functional performance, survival, quality of life and radiographic parameters of all enrolled study subjects will be evaluated in addition.

ELIGIBILITY:
Inclusion Criteria:

* Patient is capable of understanding the doctor's explanations, following his instructions and is able to participate in the follow-up program.
* Patient has given written consent to take part in the study by signing the "Patient Consent Form".
* Patient is 18-80 years of age, inclusive.
* Patient is skeletally mature.
* Patient requires a primary, fracture or revision reverse total shoulder replacement for the relief of pain and has significant disability due to gross rotator cuff deficiency.
* Patient's joint is anatomically and structurally suited to receive the selected implants.
* Patient has a functional deltoid muscle.

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patients who have any condition which would in the judgement of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, or is a known drug abuser, a known alcoholic or anyone who cannot understand what is required of them.
* Patient is known to be pregnant or breastfeeding.
* Patient is a vulnerable subject.
* Patient meets at least one of the contraindications:

  * Signs of infection
  * Significant injury to the upper brachial plexus
  * Non-functional deltoid muscle
  * Insufficient quality and/or quantity of glenoid or humeral bone
  * Any neuromuscular or vascular disease compromising the affected limb that would endanger the success of the intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe shoulder pain and disability indicated for implantation of the ASHCOM Shoulder System and who meet all inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Stamilla, MD, Principal Investigator — Clinica del Mediterraneo
Locations (1):
- Clinica del Mediterraneo, Ragusa, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: implants
Groups:
- ASHCOM Shoulder System Subjects - Uncemented Humeral Stem: Subjects implanted with the ASHCOM Shoulder System and an uncemented humeral stem.
  ASHCOM Shoulder System: Reverse Shoulder Arthroplasty
- ASHCOM Shoulder System Subjects - Fracture Humeral Stem: Subjects implanted with the ASHCOM Shoulder System and a fracture humeral stem.
  ASHCOM Shoulder System: Reverse Shoulder Arthroplasty
Period: Overall Study
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Started | 22; 22 implants | 2; 2 implants
Completed | 0; 0 implants | 0; 0 implants
Not Completed | 22; 22 implants | 2; 2 implants
Not completed — Death | 1 | 0
Not completed — Early study termination | 21 | 2

BASELINE CHARACTERISTICS:
Groups:
- ASHCOM Shoulder System Subjects - Uncemented Humeral Stem: Subjects implanted with the ASHCOM Shoulder System and an uncemented humeral stem
  ASHCOM Shoulder System: Reverse Shoulder Arthroplasty
- ASHCOM Shoulder System Subjects - Fracture Humeral Stem: Subjects implanted with the ASHCOM Shoulder System and a fracture humeral stem
  ASHCOM Shoulder System: Reverse Shoulder Arthroplasty
- Total: Total of all reporting groups
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem | Total
Number analyzed (Participants) | 22 | 2 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.14 (6.14) | 72.5 (3.54) | 70.33 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 12 | 0 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 22 | 2 | 24
Preop BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.34 (2.46) | 22.2 (1.13) | 25.99 (2.64)

OUTCOME MEASURES:

1. Primary Outcome: Survival of Implant System (Kaplan Meier)
Description: The primary endpoint is defined by the survival of the implant at 10 years which is based on removal or intended removal of the prosthesis and will be determined using Kaplan Meier method.
  Due to early study termination, the survival of the implant was analyzed at 3 years.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Number analyzed (Participants) | 21 | 2
Participants | 21 | 2

2. Secondary Outcome: The Performance and Clinical Benefits of the ASHCOM Shoulder System - Constant Murley Shoulder Score (CM)
Description: The secondary endpoint of this study is defined by the performance and clinical benefits of the ASHCOM Shoulder System at 5 years, which is assessed by the Constant and Murley score. Due to early study termination, the Constant and Murley Score was assessed at 2 years.
  The Constant and Murley score is a 100-point functional shoulder assessment tool in which higher scores reflect increased function. The subjective variables are pain (15 points) and function (activities of daily living - sleep, work, recreation/sport; 20 points), for a total of 35 points. The objective variables are active range of motion (clinician assessment; 40 points) and strength (25 points), for a total of 65 points. The minimum score is 0 points (worst outcome), the maximum score possible is 100 points (best outcome).
Time Frame: Pre-operative (baseline), 1 year, 2 years post-operative
Population: The number analyzed in one or more rows differs from overall number analyzed, as one patient passed away prior to the 3-6 month visit and for one patient the score was not collected at the 2 years follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Number analyzed (Participants) | 22 | 2
Number analyzed (Implants) | 22 | 2
score on a scale
  Preop | 7.91 (8.18) | 5.0 (7.07)
  1 year: number analyzed (Participants) | 21 | 2
  1 year: number analyzed (Implants) | 21 | 2
  1 year | 74.0 (12.55) | 55.0 (4.24)
  2 years: number analyzed (Participants) | 20 | 2
  2 years: number analyzed (Implants) | 20 | 2
  2 years | 82.95 (8.65) | 70.5 (9.19)
Statistical Analysis 1: Comparison: ASHCOM Shoulder System Subjects - Uncemented Humeral Stem; The small sample size of arm "ASHCOM Shoulder System subjects - Fracture humeral stem" of 2 cases is too low for a statistical analysis; Test type: Other — P-values account for preoperative versus postoperative mean values at 1 and 2 years; p < .0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Oxford Shoulder Score (OSS)
Description: The Oxford Shoulder Score (OSS) is a patient-reported outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following total shoulder arthroplasty. The OSS consists of twelve questions covering function and pain associated with the shoulder. To calculate the total score, each question is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible and a minimum of 0, representing the worst possible.
  The outcome score can be categorized as: Satisfactory Joint Function: 40 - 48, Moderate-Mild Arthritis: 30 - 39, Moderate-Severe Arthritis: 20 - 29, Severe Arthritis: 0 - 19.
Time Frame: Pre-operative (baseline), 3-6 months, 1 year, 2 and 3 years post-operative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Number analyzed (Participants) | 22 | 2
Number analyzed (Implants) | 22 | 2
score on a scale
  Preop | 6.27 (3.56) | 5.5 (7.78)
  3-6 Month: number analyzed (Participants) | 21 | 2
  3-6 Month: number analyzed (Implants) | 21 | 2
  3-6 Month | 41.81 (3.97) | 32.5 (0.71)
  1 Year: number analyzed (Participants) | 21 | 2
  1 Year: number analyzed (Implants) | 21 | 2
  1 Year | 47.62 (0.92) | 45.5 (0.71)
  2 Year: number analyzed (Participants) | 20 | 2
  2 Year: number analyzed (Implants) | 20 | 2
  2 Year | 47.8 (0.52) | 48.0 (0.0)
  3 Year: number analyzed (Participants) | 21 | 2
  3 Year: number analyzed (Implants) | 21 | 2
  3 Year | 48.0 (0.0) | 47.5 (0.71)
Statistical Analysis 1: Comparison: ASHCOM Shoulder System Subjects - Uncemented Humeral Stem; [analysis description as in outcome 2, analysis 1]; Test type: Other — P-values account for preoperative versus postoperative mean values at 3-6 months, 1 year, 2 and 3 years; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: EQ-5D-5L Score
Description: The EQ-5D-5L is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, self-care, daily activities, pain/discomfort and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. In the derived EQ-5D-5L score, the highest score is 1 and the lowest score is -0.573. It included the Health State, which is a self-reported assessment about the patient's health on that day at a VAS from 0 to 100 with 100 being the best health one can imagine and 0 the worst.
Time Frame: Pre-operative (baseline), 3-6 months, 1 year, 2 and 3 years post-operative
Population: The number analyzed in one or more rows differs from overall number analyzed, as one patient passed away prior to the 3-6 month visit and for one patient the score was not collected at the 3-6 months and 1 year follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Number analyzed (Participants) | 22 | 2
score on a scale
  Preop | 0.22 (0.16) | 0.06 (0.07)
  3-6 Months: number analyzed (Participants) | 20 | 2
  3-6 Months | 0.79 (0.11) | 0.56 (0.15)
  1 Year: number analyzed (Participants) | 20 | 2
  1 Year | 0.97 (0.08) | 0.67 (0.17)
  2 Year: number analyzed (Participants) | 21 | 2
  2 Year | 0.99 (0.05) | 0.88 (0.0)
  3 Year: number analyzed (Participants) | 21 | 2
  3 Year | 1.0 (0.01) | 0.97 (0.04)
Statistical Analysis 1: Comparison: ASHCOM Shoulder System Subjects - Uncemented Humeral Stem; [analysis description as in outcome 2, analysis 1]; Test type: Other — P-values account for preoperative versus postoperative mean values at 3-6 months, 1, 2 and 3 years; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Subjective Shoulder Value (SSV)
Description: The Subjective Shoulder Value (SSV) is a single point, subjective estimate of a patient's condition. The patient is asked to rate the functionality of their operated shoulder on a scale of 0% - 100% of normal.
Time Frame: Pre-operative (baseline), 3-6 months, 1 year, 2 and 3 years post-operative
Population: The number analyzed in one or more rows differs from overall number analyzed, as one patient passed away prior to the 3-6 month visit. For one patient the score was not collected at the 3-6 months follow-up visit and for two patients at the 1 year follow-up visit.
Measure: Mean (Standard Deviation); unit: percentage of normal
Units Other Than Participants: Implants
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Number analyzed (Participants) | 22 | 2
Number analyzed (Implants) | 22 | 2
percentage of normal
  Preop | 25.0 (14.72) | 10.0 (14.14)
  3-6 Months: number analyzed (Participants) | 20 | 2
  3-6 Months: number analyzed (Implants) | 20 | 2
  3-6 Months | 76.5 (9.47) | 62.5 (3.54)
  1 Year: number analyzed (Participants) | 19 | 2
  1 Year: number analyzed (Implants) | 19 | 2
  1 Year | 89.74 (9.64) | 77.5 (3.54)
  2 Year: number analyzed (Participants) | 19 | 2
  2 Year: number analyzed (Implants) | 19 | 2
  2 Year | 94.74 (7.35) | 90.0 (0.0)
  3 Year: number analyzed (Participants) | 21 | 2
  3 Year: number analyzed (Implants) | 21 | 2
  3 Year | 96.19 (5.46) | 97.5 (3.54)
Statistical Analysis 1: Comparison: ASHCOM Shoulder System Subjects - Uncemented Humeral Stem; [analysis description as in outcome 2, analysis 1]; Test type: Other — P-values account for preoperative versus postoperative mean values at 3-6 months, 1 year, 2 and 3 years; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Radiographic Parameters
Description: Radiographic parameters: X-rays have been evaluated for radiolucency, osteolysis, atrophy, hypertrophy, osteophytes (glenoid), component migration (humeral stem subsidence / glenoid component migration), heterotopic ossification and scapular notching
Time Frame: 2 years post-operative
Population: ASHCOM Shoulder System subjects - Uncemented humeral stem: The number analyzed at 2 years is 21, as one patient passed away prior to the 3-6 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
Number analyzed (Participants) | 21 | 2
Participants
  Any radiographic findings - Yes: | 0 | 0
  Any radiographic findings - No: | 21 | 2

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of surgery until study termination (up to 3 years)
Arm/Group | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem | ASHCOM Shoulder System Subjects - Fracture Humeral Stem
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/2
Other Adverse Events (participants affected / at risk) | 0/22 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASHCOM Shoulder System Subjects - Uncemented Humeral Stem (N=22) | ASHCOM Shoulder System Subjects - Fracture Humeral Stem (N=2)
Not study related death (General disorders) | 1 (1) | 0 (0) — Patient died from Covid two months after surgery

LIMITATIONS AND CAVEATS:
Limitations of this study are the low overall sample size of 24 cases as well as the short follow-up period of three years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT04258605/Prot_SAP_000.pdf